CLINICAL TRIAL: NCT03744949
Title: Determination of the ED50 and ED95 of Remifentanil to Perform Tracheal Intubation Without Significant NOL Index Variation
Brief Title: ED50 and ED95 of Remifentanil for Intubation Without NOL Variation
Acronym: RemiTrach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Director of Research in the Department of Anesthesiology, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-1410
Record Dates: First submitted 2018-11-11; First posted 2018-11-19 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Intubation; Difficult or Failed
Keywords: Tracheal intubation; Remifentanil; Pain; NOL index; Anesthesia; Analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Four groups of patients. Randomization into the dose of remifentanil given according to a randomization list for a total number of patients of 80.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: remifentanil will be given by a dosage of 0.5-1.0-1.5-2.0 µg/kg of adjusted body weight bolus according to randomization, by an infusion pump over 30 seconds
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Remifentanil dose 0.5 ug/kg (Experimental): Remifentanil will be given (dosage of 0.5 µg/kg of adjusted body weight bolus) from an infusion pump over 30 seconds. The bolus of remifentanil will be programmed on an electronic pump which gives an auditory signal when each bolus is completed. When the pump will ring at the end of the remifentanil bolus, the chronometer on the Dräger Monitor (anesthesia machine, Dräger Perseus A500, Draeger Medical Canada Inc., Ontario, Canada) will be turned on.
  Interventions: Drug: Remifentanil dose 0.5 ug/kg
- Remifentnil dose 1 ug/kg (Experimental): Remifentanil will be given (dosage of 1.0 µg/kg of adjusted body weight bolus according to randomization) from an infusion pump over 30 seconds. The bolus of remifentanil will be programmed on an electronic pump which gives an auditory signal when each bolus is completed. When the pump will ring at the end of the remifentanil bolus, the chronometer on the Dräger Monitor (anesthesia machine, Dräger Perseus A500, Draeger Medical Canada Inc., Ontario, Canada) will be turned on.
  Interventions: Drug: Remifentanil dose 1 ug/kg
- Remifentanil dose 1.5 ug/kg (Experimental): Remifentanil will be given (dosage of 1.5 µg/kg of adjusted body weight bolus according to randomization) from an infusion pump over 30 seconds. The bolus of remifentanil will be programmed on an electronic pump which gives an auditory signal when each bolus is completed. When the pump will ring at the end of the remifentanil bolus, the chronometer on the Dräger Monitor (anesthesia machine, Dräger Perseus A500, Draeger Medical Canada Inc., Ontario, Canada) will be turned on.
  Interventions: Drug: Remifentanil dose 1.5 ug/kg
- Remifentanil dose 2 ug/kg (Experimental): Remifentanil will be given (dosage of 2 µg/kg of adjusted body weight bolus according to randomization) from an infusion pump over 30 seconds. The bolus of remifentanil will be programmed on an electronic pump which gives an auditory signal when each bolus is completed. When the pump will ring at the end of the remifentanil bolus, the chronometer on the Dräger Monitor (anesthesia machine, Dräger Perseus A500, Draeger Medical Canada Inc., Ontario, Canada) will be turned on.
  Interventions: Drug: Remifentanil dose 2 ug/kg

INTERVENTIONS:
Drug: Remifentanil dose 0.5 ug/kg — Remifentanil will be given (dosage of 0.5 µg/kg of adjusted body weight bolus) from an infusion pump over 30 seconds
  Arms: Remifentanil dose 0.5 ug/kg
Drug: Remifentanil dose 1 ug/kg — Remifentanil will be given (dosage of 1 µg/kg of adjusted body weight bolus) from an infusion pump over 30 seconds
  Arms: Remifentnil dose 1 ug/kg
Drug: Remifentanil dose 1.5 ug/kg — Remifentanil will be given (dosage of 1.5 µg/kg of adjusted body weight bolus) from an infusion pump over 30 seconds
  Arms: Remifentanil dose 1.5 ug/kg
Drug: Remifentanil dose 2 ug/kg — Remifentanil will be given (dosage of 2 µg/kg of adjusted body weight bolus) from an infusion pump over 30 seconds
  Arms: Remifentanil dose 2 ug/kg

SUMMARY:
Our aim, in this study, is to elucidate the optimal dosing range (ED50 and ED95) of bolus remifentanil in order to counter the painful stimuli resulting from direct laryngoscopy and tracheal intubation by using the NOL index. In order to maximize the clinical relevance of our findings, induction of general anesthesia will be done with standard medications and doses and laryngoscopy will be done with the Macintosh laryngoscope, the most common tool used for intubation in the operating room

DETAILED DESCRIPTION:
Background: There are no study so far that determined the ED50 and ED95 of remifentanil to perform tracheal intubation by using the NOL index as the criterion measured to determine the failure (painful intubation) or the success (pain free intubation) of the assessed procedure.

Objectives: To determine the ED50 and ED95 of remifentanil bolus to perform tracheal intubation without NOL index variating over threshold for nociceptive response (determined as a NOL index going over 20 - peak value of maximum 20) using the Macintosh blade when obtaining good conditions of intubation in anesthetized patients. Good conditions of intubation will be determined as obtaining a Cormack-Lehane grade I and II.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I or II
* Mallampati class I or II
* Patients > 18 years old and <65 years (defining elderly patients)
* Elective general, gynecological, orthopedic, plastic or urological surgery under general anesthesia
* Type of surgery that usually necessitate endotracheal intubation and controlled ventilation

Exclusion Criteria:

* Patient refusal
* History of psychiatric diseases or psychological problems (including mental retardation); inability to give consent; language barrier.
* Anticipated difficult airway (Mallampati class III and IV, thyromental distance < 6 cm, mouth opening < 3 cm, neck extension <80° and neck flexion <35°, inability to prognath, meaning bringing lower mandibular before the upper maxilla)
* Patient with history of neck rigidity or instability
* BMI > 30 kg/m2
* Anticipated difficult ventilation (patients with beard, obesity with BMI more than 30 kg/m2)
* Patient with history of oropharyngeal or tracheal surgery (excluding adenoidectomy, tonsillectomy and teeth removal)
* Severe coronary artery disease
* Serious cardiac arrhythmias (including atrial fibrillation)
* Use of β-blockers (all types)
* History of opioid or illicit drug substance abuse
* Chronic use of psychotropic and/or opioid drugs
* Allergy to remifentanil or propofol
* Pregnancy
* Contraindications to mask ventilation (gastrointestinal tract obstruction, pregnancy, active not-treated gastroesophageal reflux disease, non-fasting patients)
* Unexpected difficult airway requesting excessive, possibly painful airway manipulations
* Requiring hemodynamic support with vasopressors or inotropes 2 min before laryngoscopy to 5 min after insertion of endotracheal tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
determine ED95 of remifentanil bolus in mcg/kg for tracheal intubation | in the surgery
  The primary goal of this study is to determine the ED95 of remifentanil bolus to perform tracheal intubation without NOL index varying over 20 (peak maximal value of 20) using the Macintosh blade when obtaining a Cormack-Lehane grade I or II of intubation in anesthetized patients (the size of the blade will be chosen according to patient characteristics described in the user's manual for each blade and published in previous literature). This primary outcome will be expressed in mcg/kg of remifentanil.

SECONDARY OUTCOMES:
NOL maximal value after intubation (NOL is an index without unit going from 0 to 100) | in the surgery
  After tracheal intubation NOL index maximal value will be evaluated and compared between the 4 doses of remifentanil in mcg/kg received in this study.
Variation of NOL index after tracheal intubation; DELTA NOL (no unit) | in the surgery
  After tracheal intubation DELTA NOL index will be evaluated and compared between the 4 doses of remifentanil in mcg/kg received in this study.
Time in seconds NOL spends above 25 after tracheal intubation (in seconds) | in the surgery
  Time in seconds spent above 25 of NOL index and comparison between the 4 doses of remifentanil used in this study
Area under the curve for NOL index after tracheal intubation (no unit) | in the surgery
  Compare the AUC of NOL after tracheal intubation between the 4 doses of remifentanil used in this study.
Heart Rate Maximal value after tracheal intubation (in beat per minutes) | in the surgery
  To compare maximal heart rate values reached after tracheal intubation between the 4 doses of remifentanil used in this study
Heart Rate variation (DELTA Heart Rate) after tracheal intubation (in beats per minute) | in the surgery
  To compare the DELTA Heart Rate after tracheal intubation between the 4 doses of remifentanil used in this study
Time in seconds that Heart Rate spends above threshold of 10%; in seconds | in the surgery
  To compare the time in seconds between the 4 doses of remifentanil that Heart Rate spends above teh threshold of 10% of variation above normal prestimulus values.
Area under the curve of Heart Rate after tracheal intubation (no unit) | in the surgery
  To compare AUC of Heart Rate values after tracheal intubation between teh 4 different doses of remifentanil used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebe, MD PhD, Principal Investigator — CIUSSS de l'Est de Montreal, Hopital Maisonneuve Rosemont
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No